CLINICAL TRIAL: NCT03099564
Title: A Pilot Study of Pembrolizumab in Combination With Y90 Radioembolization in Subjects With Poor Prognosis Hepatocellular Carcinoma With Preserved Liver Function. HCRN: GI15-225
Brief Title: Pembrolizumab Plus Y90 Radioembolization in HCC Subjects
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ashwin Somasundaram (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Ashwin Somasundaram, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GI15-225
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Pembrolizumab; Y90 Radioembolization; KEYTRUDA®; TheraSphere®; PD-1; IgG4/kappa isotype
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- pembrolizumab + Y90 radioembolization (Experimental): Pembrolizumab 200mg IV every 3 weeks in conjunction with Y90 radioembolization (performed one week after the first dose of pembrolizumab)
  Interventions: Drug: Pembrolizumab; Device: Y90 radioembolization

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab 200mg IV every three weeks
  Other Names: Keytruda®
Device: Y90 radioembolization — The first Y90 radioembolization treatment will be administered one week after the first dose of pembrolizumab. If a second Y90 radioembolization treatment is required for bilobar disease, this should occur within 4 weeks of the initial procedure (between Cycles 2 and 3 of pembrolizumab).

SUMMARY:
This is an open-label multi-center trial designed to evaluate the efficacy as well as the safety of combining pembrolizumab with Yttrium-90 (Y90) radioembolization in subjects with poor prognosis (high risk) HCC not eligible for liver transplant or surgical resection with well compensated liver function. Treatment will consist of pembrolizumab 200mg IV every 3 weeks in conjunction with Y90 radioembolization performed one week after the first dose of pembrolizumab. If bilobar disease is present, a second Y90 radioembolization will be performed no later than 4 weeks after the first procedure to the contralateral hepatic lobe.

DETAILED DESCRIPTION:
If a second Y90 radioembolization treatment is required for bilobar disease, this should occur within 4 weeks of the initial procedure (between Cycles 2 and 3 of pembrolizumab). The next dose of pembrolizumab should be separated from the Y90 radioembolization by at least one week.

Imaging will be obtained every 9 weeks (after every 3 pembrolizumab treatment) to assess for tumor response and to evaluate for progression. Subjects will remain on treatment until documented tumor progression, unacceptable toxicity, study withdrawal or death.

Screening Angiography (shunt study):

During screening, subjects will undergo angiography using technetium-99-labeled macroaggregated albumin to detect any uptake outside the liver via measurement of hepatopulmonary shunting. Prior to the angiography, a local anesthetic (to numb the area prior to catheter insertion) and sedation will be administered to the subject, as per institutional standards.

This procedure is standard of care for subjects prior to Y90 radioembolization, and will be performed per institutional site standards. Hepatopulmonary shunting must be < 20% for subject to meet eligibility criteria. Subjects will undergo a mandatory tumor biopsy on the same day as the screening angiography.

Prior to administration of the first dose of pembrolizumab (i.e., Day 1 of Cycle 1), repeat laboratory tests will be obtained to ensure subject still meets eligibility criteria.

Pembrolizumab 200mg IV (IV over 30 minutes) every 3 weeks Day 1 per 21 day cycle (3 weeks).

Prior to administration of subsequent pembrolizumab doses, the following criteria must be met:

ALT and AST:

* Among subjects with baseline (screening) ALT/AST <2×ULN: ALT/AST < 5×ULN
* Among subjects with baseline (screening) ALT/AST ≥2×ULN: ALT/AST < 3× the baseline level
* ALT/AST ≤ 500 U/L regardless of baseline level

Total bilirubin:

* Among subjects with baseline levels < 1.5 mg/dL: a value of < 2.0 mg/dL
* Among subjects with baseline levels that are ≥ 1.5 mg/dL: a value < 2× the baseline level
* Total bilirubin ≤ 3.0 mg/dL regardless of baseline level

Y90 radioembolization will be performed as standard of care via institutional standards.

To be eligible for Y90 radioembolization, the following criteria must be met:

ALT and AST:

* Among subjects with baseline (screening) ALT/AST < 2×ULN: ALT/AST < 5×ULN
* Among subjects with baseline (screening) ALT/AST ≥ 2×ULN: ALT/AST < 3× the baseline level
* ALT/AST ≤ 500 U/L regardless of baseline level

Total bilirubin:

* Among subjects with baseline levels < 1.5 mg/dL: a value of < 2.0 mg/dL
* Among subjects with baseline levels that are ≥ 1.5 mg/dL: a value < 2× the baseline level
* Total bilirubin ≤ 3.0 mg/dL regardless of baseline level

In addition, any non-hepatic toxicities from the prior dose(s) of pembrolizumab must have resolved to Grade ≤ 2.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately
* ECOG Performance Status of 0-1
* Locally advanced HCC as defined by: 1) tissue diagnosis OR 2) alpha-fetoprotein (AFP) > 400 ng/mL with compatible mass on contrast-enhanced imaging OR 3) compatible mass on dual phase CT or dynamic contrast enhanced MRI demonstrating both arterial hypervascularity and delayed washout
* Hepatopulmonary shunting < 20% as documented via hepatic artery perfusion study
* No evidence of extrahepatic metastatic disease
* Subjects must be considered poor prognosis by the following parameters: 1) right or left portal vein involvement (NOTE: subjects with main portal vein involvement are excluded), 2) multi-focal disease (more than 3 tumors regardless of size) AND/OR 3) diffuse disease considered amenable to liver directed therapy.
* Subjects with chronic infection by HCV who are untreated or who failed previous therapies for HCV are allowed on study. In addition, subjects with successful HCV treatment (defined as sustained virologic response [SVR] 12 or SVR 24) are allowed as long as patients are not actively receiving anti-HCV treatment at the time of study enrollment. Investigators can stop anti-HCV treatment at their discretion prior to enrolling patients on study. .
* If active HBV, viral load must be <100IU/mL; if active HBV, subjects must be on anti-viral medication for ≥ 3 months prior to study registration and remain on the same anti-viral regimen throughout study treatment. NOTE: those subjects who are positive for Hepatitis B core antibody (anti-HBc), negative for Hepatitis B surface antigen (HBsAg) and negative for Hepatitis B surface antibody (anti-HBs), and have an HBV viral load <100 IU/mL do not require HBV anti-viral prophylaxis.
* Not eligible for surgical resection or liver transplant or have refused such procedures.
* All disease must be amenable to embolization in one or two procedures
* Childs-Pugh Cirrhotic Status A or B with a maximum score of 7
* No evidence of clinically apparent ascites or active encephalopathy, and/or varices that have not been treated. Subjects with controlled ascites or encephalopathy are eligible so long as they meet Childs-Pugh score criterion. Please note that controlled ascites and encephalopathy require scores of 2 each when calculating the C-P score.
* No prior systemic therapy or radiotherapy (including Y90 radioembolization or cyberknife) for HCC. No prior TAE or TACE allowed. Previous liver resection and ablation therapy is permitted. Allowed prior therapies must be completed 4 weeks prior to the baseline scan, and untreated measurable disease (as per RECIST1.1) must be present.
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to registration:

Hematological:

Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L; Hemoglobin (Hgb) ≥ 9 g/dL; Platelet Count ≥ 60 x 10^9/L

Renal:

Calculated creatinine clearance ≥ 60 cc/min

Hepatic:

Bilirubin < 2.0 X ULN; Aspartate aminotransferase (AST) ≤ 5 × ULN; Alanine aminotransferase (ALT) ≤ 5 × ULN

Coagulation:

International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5

* Females of childbearing potential must have a negative serum pregnancy test within 72 hours prior to registration.
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use effective methods of contraception from the time of informed consent until 120 days after treatment discontinuation.
* Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study
* Is willing to undergo a mandatory pre-treatment (all subjects) and post-treatment (10 subjects) research biopsy at the centers participating in research biopsies

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of study registration
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy (other than oral contraceptives) or any other form of immunosuppressive therapy within 7 days prior to registration.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g.thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency.) is not considered a form of systemic treatment.
* Known history of active TB
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to registration or who has not recovered (i.e., ≤ Grade 1 or baseline) from adverse events due to agents administered > 4 weeks prior
* Has had prior chemotherapy, targeted small molecule therapy or radiation therapy within 2 weeks prior to registration, or who has not recovered (i.e., (i.e., ≤ Grade 1 or baseline)) from AEs due to previously administered agents
* If had major surgery, subject must have recovered adequately from the toxicity and/or complications from the intervention prior to study registration
* Complete portal vein occlusion
* Vascular abnormalities or bleeding diathesis that indicates hepatic artery catheterization is contraindicated
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody
* Known history of HIV
* Untreated active HBV
* Dual infection with HBV/HCV or other hepatitis combinations at study entry
* Known history of, or any evidence of active, non-infectious pneumonitis
* History of organ or stem cell transplantation including previous history of liver transplantation
* Active infection requiring systemic therapy
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Has history or current evidence of any condition, therapy or laboratory abnormality that may confound results or interfere with subject's participation in the trial.
* Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least three years.
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 months
  Freedom from progression or death at 6 months based on RECIST 1.1 criteria

SECONDARY OUTCOMES:
Assess Safety - toxicities as defined by the NCI CTCAE v4 | 2 years
  Grade 3 and 4 toxicities as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v4
Time to progression (TTP) | 2 years
  Time from Day 1 (D1) of pembrolizumab to progression
Objective response rate (ORR) | 2 years
  Per RECIST1.1 and mRECIST for Hepatocellular Carcinoma (HCC) and will be calculated as the number of subjects with a Complete Response (CR) or Partial Response (PR) divided by the total number of evaluable subjects
Estimate overall survival (OS) | 3 years
  The time from Day 1 (D1) of pembrolizumab to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Somasundaram, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Washington/Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Yu S, Yu M, Keane B, Mauro DM, Helft PR, Harris WP, Sanoff HK, Johnson MS, O'Neil B, McRee AJ, Somasundaram A. A Pilot Study of Pembrolizumab in Combination With Y90 Radioembolization in Subjects With Poor Prognosis Hepatocellular Carcinoma. Oncologist. 2024 Mar 4;29(3):270-e413. doi: 10.1093/oncolo/oyad331. PMID 38325328
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org